CLINICAL TRIAL: NCT04252794
Title: Graft Inflow Modulation for Portal Hyper-perfusion in Live Donor Liver Transplantation: a Randomized Pilot Study
Brief Title: Graft Inflow Modulation for Portal Hyper-perfusion in Live Donor Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Principal Investigator, Gattu Tharun, Senior Resident, HPB Surgery, Institute of Liver and Biliary Sciences, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILBS-Liver Transplant-02
Record Dates: First submitted 2020-01-10; First posted 2020-02-05 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who undergo GIM (Experimental): If inclusion criteria are met, after randomisation, these group of patients will undergo splenic artery ligation (graft inflow modulation)
  Interventions: Procedure: Splenic artery ligation
- No splenic artery ligation (Active Comparator): If inclusion criteria are met, after randomisation, these group of patients will not undergo splenic artery ligation (graft inflow modulation)
  Interventions: Other: No intervention

INTERVENTIONS:
Procedure: Splenic artery ligation — Splenic artery will be ligated just after takeoff from coeliac trunk at the level of body of pancreas
  Arms: Patients who undergo GIM
Other: No intervention — Splenic artery is not ligated despite the presence of portal hyperperfusion
  Arms: No splenic artery ligation

SUMMARY:
In this study, the investigators aim to prove that performing graft inflow modulation (GIM) in liver with portal hyper-perfusion is beneficial for early graft function postoperatively. Grafts at risk for portal hyper-perfusion will be identified by doing an intraoperative Doppler after reperfusion. In group A, the investigators will take 21 liver transplant recipients after reperfusion, randomly allocated, who will undergo intraoperative graft inflow modulation by splenic artery ligation. In group B, the investigators will be analyzing another randomly allocated 21 patients, who will not undergo any graft inflow modulation. The investigators will be analyzing trend of LFT's (liver function tests) after surgery, time for normalization of bilirubin, INR (international normalised ratio) and decrease in ascites, morbidity, mortality, ICU (intensive care unit) and total hospital stay.

DETAILED DESCRIPTION:
Due to shortage of deceased donor organs, LDLT (living donor living transplantation) is gaining importance all over world. Previous studies have showed poor outcomes with donor grafts having GRWR (graft to recipient weight ratio) < 0.8 due to development of SFSS (Small for Size Syndrome) where the graft is too small to meet the recipient's metabolic demands. SFSS is characterised by prolonged cholestasis, intractable ascites, prolonged INR and encephalopathy. However, it is not always possible to obtain larger graft from live donor owing to the risk's associated to donor. Various techniques have been developed in order to manage a smaller graft in recipient (ex: hemiportocaval shunts, splenic artery ligation, splenectomy). HPCS (hemiportocaval shunt) have been associated with risks of portal steal phenomenon and encephalopathy. Splenectomy is associated with increased risks of infections / sepsis and portal vein thrombosis postoperatively. Splenic artery ligation close to its origin is associated with least risks and is increasingly being used as the method of graft inflow modulation when required.

Recent studies have showed that Portal Flow Hemodynamics are more important than GRWR in predicting the occurrence of SFSS. Grafts whose GRWR is > 0.8 can also show features of SFSS after ruling out all other causes (5). Persistent portal hypertension leads to sinusoidal endothelial injury, haemorrhage, oedema and architectural distortion - these changes are more marked in SFS (small for size) grafts. Also, due to hepatic arterial buffer response, reduced flow in hepatic artery leads to further ischemic injury, cholestasis and ischemic cholangitis. A recipient portal venous flow of > 250 ml/min/100 grams of liver weight is defined as portal hyper perfusion.

H Y Ou et al retrospectively analysed data involving patients whose PVF > 250 ml/min/100 gr after reperfusion where 6 patients underwent inflow modulation (using splenic artery ligation) and other 2 didn't. They found that only 1 / 6 patients in those who underwent GIM developed SFSS where as both the patients who didn't undergo GIM developed SFSS (1 of them died). Also, none of the patients developed complications related to splenic artery ligation in their study.

Bhavin B et al in their retrospective study on 134 liver transplant recipients found that 19 patients met criteria for SFSS (as per Kyushu University). On analysis of the factors responsible for early graft dysfunction, only portal vein flow > 190 ml/min/100 gr of liver after reperfusion was found to be a significant predictor. GRWR was not significantly associated with graft dysfunction - 3 / 19 patients had GRWR < 0.8 while 16 patients in non-dysfunction group had GRWR < 0.8

Ogura et al retrospectively analysed data involving intentional portal pressure modulation when PVP (portal venous pressure) > 20 mm Hg. They found that the patients with a portal pressure < 15 mm Hg had better 2 year survival compared to those with > 15 mm Hg. Also, recovery from hyper bilirubinaemia and coagulopathy after transplantation was significantly better in those with PVP < 15 mm Hg.

Wang et al retrospectively analysed data involving 276 patients where they performed GIM by doing splenectomy (SPL) when PVP > 20 mm Hg. Group 1 had 134 patients who underwent SPL and Group 2 had 122 patients in whom GIM was not done. Graft compliance, Portal venous flow was significantly better in group 1 patients. Also, there was faster normalisation of bilirubin and ascites in group 1 when compared to group 2. Overall, 15.6 % patients had complications related to SPL - bleeding from splenic hilum, pancreatic leak, OPSS (overwhelming post spleenectomy sepsis) (1.9%).

Luca A et al in their study involving cirrhotic patients with portal hypertension, splenic artery occlusion causes a significant reduction in portal pressure gradient (PPG). This drop was indirectly related to liver volume and directly related to spleen volume. The spleen/liver volume ratio> 0.5 accurately predicts the drop in PPG and may be used to identify patients who can obtain a significant advantage from procedures decreasing splenic inflow.

Ayman et al had done a study wherethey aimed to keep final PVP < 20 mm Hg and analysed if PVP > 15 is a better predictor than PVP > 20 mm Hg for SFSS. Peak bilirubin, INR, incidence of post-transplant HE and SFSS was significantly higher in those with PVP of 15 - 19 mm Hg (group B) vs in those with PVP < 15 mm Hg (group A). 90 day morbidity and mortality was also significantly higher in Group B when compared to group A. On comparing grafts with GRWR < 0.8 with > 0.8, no significant differences in postoperative outcomes were seen.

Troisi et al did a retrospective study where they used Splenic artery ligation as the method of GIM when Recipient Portal Venous Flow was three times that of Donor portal vein flow. Group 1 had 11 patients with no GIM and group 2 had 13 patients who underwent GIM. SFSS occurred in three patients in Group 1 where all three needed re-transplantation whereas none of the patients in Group 2 developed SFSS. Also, One-year overallsurvival was 62% and 93% respectively for Group 1 and Group 2.

ELIGIBILITY:
Inclusion Criteria:

* Portal Venous Pressure (PVP) > 15 mm Hg after reperfusion or
* Portal venous flow (PVF) > 250 ml/min/100 gr of liver after reperfusion with a gradient (PVP - CVP) of ≥ 7 mm Hg

Exclusion Criteria:

* Significant peripancreatic collaterals preventing safe access to splenic artery
* Acute Liver Failure as an indication for transplant
* ABO incompatible transplants
* Pediatric transplants
* Refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of early graft dysfunction | first postoperative month
  Number of patients who develop early graft dysfunction in each group

SECONDARY OUTCOMES:
Time to normalisation of bilirubin | first postoperative month
  time to normalisation of bilirubin (in days)
Time to normalisation of INR | first postoperative month
  time to normalisation of INR (in days)
Time to normalisation of ascites output | first postoperative month
  time to normalisation of ascites output (in days)
Morbidity | first postoperative month
  Morbidity as per Clavein Dindo classfification
ICU stay | first operative month
  Duration of ICU stay (in days)
Mortality | first postoperative month
  death
Total hospital stay | till 3 months after surgery
  duration of total stay in hospital after liver transplatation (in days)

CONTACTS AND LOCATIONS:
Overall Officials: Gattu Tharun, MS, Principal Investigator — Senior resident, Department of HPB surgery, ILBS, India
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kiuchi T, Kasahara M, Uryuhara K, Inomata Y, Uemoto S, Asonuma K, Egawa H, Fujita S, Hayashi M, Tanaka K. Impact of graft size mismatching on graft prognosis in liver transplantation from living donors. Transplantation. 1999 Jan 27;67(2):321-7. doi: 10.1097/00007890-199901270-00024. PMID 10075602
- [Result] Bell R, Pandanaboyana S, Upasani V, Prasad R. Impact of graft-to-recipient weight ratio on small-for-size syndrome following living donor liver transplantation. ANZ J Surg. 2018 May;88(5):415-420. doi: 10.1111/ans.14245. PMID 29752783
- [Result] Vasavada BB, Chen CL, Zakaria M. Portal flow is the main predictor of early graft dysfunction regardless of the GRWR status in living donor liver transplantation - a retrospective analysis of 134 patients. Int J Surg. 2014;12(2):177-80. doi: 10.1016/j.ijsu.2013.12.006. Epub 2013 Dec 25. PMID 24370677
- [Result] Vasavada B, Chen CL, Zakaria M. Using low graft/recipient's body weight ratio graft with portal flow modulation an effective way to prevent small-for-size syndrome in living-donor liver transplant: a retrospective analysis. Exp Clin Transplant. 2014 Oct;12(5):437-42. PMID 25299370
- [Result] Lei JY, Yan LN, Li B, Wen TF, Wang WT, Xu MQ, Yang JY. Graft size alone should not affect donors selection and be used to predict the prognosis of recipients after living donor liver transplantation. Hepatogastroenterology. 2012 Jan-Feb;59(113):224-7. doi: 10.5754/hge11035. PMID 22260833
- [Result] Demetris AJ, Kelly DM, Eghtesad B, Fontes P, Wallis Marsh J, Tom K, Tan HP, Shaw-Stiffel T, Boig L, Novelli P, Planinsic R, Fung JJ, Marcos A. Pathophysiologic observations and histopathologic recognition of the portal hyperperfusion or small-for-size syndrome. Am J Surg Pathol. 2006 Aug;30(8):986-93. doi: 10.1097/00000478-200608000-00009. PMID 16861970
- [Result] Shimamura T, Taniguchi M, Jin MB, Suzuki T, Matsushita M, Furukawa H, Todo S. Excessive portal venous inflow as a cause of allograft dysfunction in small-for-size living donor liver transplantation. Transplant Proc. 2001 Feb-Mar;33(1-2):1331. doi: 10.1016/s0041-1345(00)02496-9. No abstract available. PMID 11267312
- [Result] Ou HY, Huang TL, Chen TY, Tsang LL, Chen CL, Cheng YF. Early modulation of portal graft inflow in adult living donor liver transplant recipients with high portal inflow detected by intraoperative color Doppler ultrasound. Transplant Proc. 2010 Apr;42(3):876-8. doi: 10.1016/j.transproceed.2010.02.064. PMID 20430194
- [Result] Ogura Y, Hori T, El Moghazy WM, Yoshizawa A, Oike F, Mori A, Kaido T, Takada Y, Uemoto S. Portal pressure <15 mm Hg is a key for successful adult living donor liver transplantation utilizing smaller grafts than before. Liver Transpl. 2010 Jun;16(6):718-28. doi: 10.1002/lt.22059. PMID 20517905
- [Result] Wang H, Ikegami T, Harada N, Yoshizumi T, Soejima Y, Uchiyama H, Yamashita Y, Itoh S, Harimoto N, Kawanaka H, Shirabe K, Maehara Y. Optimal changes in portal hemodynamics induced by splenectomy during living donor liver transplantation. Surg Today. 2015 Aug;45(8):979-85. doi: 10.1007/s00595-014-0999-9. Epub 2014 Aug 2. PMID 25080864
- [Result] Luca A, Miraglia R, Caruso S, Milazzo M, Gidelli B, Bosch J. Effects of splenic artery occlusion on portal pressure in patients with cirrhosis and portal hypertension. Liver Transpl. 2006 Aug;12(8):1237-43. doi: 10.1002/lt.20762. PMID 16741929
- [Result] Osman AM, Hosny AA, El-Shazli MA, Uemoto S, Abdelaziz O, Helmy AS. A portal pressure cut-off of 15 versus a cut-off of 20 for prevention of small-for-size syndrome in liver transplantation: A comparative study. Hepatol Res. 2017 Mar;47(4):293-302. doi: 10.1111/hepr.12727. Epub 2016 May 11. PMID 27084787
- [Result] Troisi R, de Hemptinne B. Clinical relevance of adapting portal vein flow in living donor liver transplantation in adult patients. Liver Transpl. 2003 Sep;9(9):S36-41. doi: 10.1053/jlts.2003.50200. PMID 12942477
- [Result] Yamada T, Tanaka K, Uryuhara K, Ito K, Takada Y, Uemoto S. Selective hemi-portocaval shunt based on portal vein pressure for small-for-size graft in adult living donor liver transplantation. Am J Transplant. 2008 Apr;8(4):847-53. doi: 10.1111/j.1600-6143.2007.02144.x. Epub 2008 Feb 5. PMID 18261170
- [Result] Umeda Y, Yagi T, Sadamori H, Matsukawa H, Matsuda H, Shinoura S, Mizuno K, Yoshida R, Iwamoto T, Satoh D, Tanaka N. Effects of prophylactic splenic artery modulation on portal overperfusion and liver regeneration in small-for-size graft. Transplantation. 2008 Sep 15;86(5):673-80. doi: 10.1097/TP.0b013e318181e02d. PMID 18791439
- See also: Hemodynamic interaction between portal vien and hepatic artery flow in small-for-size split liver transplantation - Smyrniotis - 2002 - Transplant International - Wiley Online Library — http://onlinelibrary.wiley.com/doi/abs/10.1111/j.1432-2277.2002.tb00178.x